CLINICAL TRIAL: NCT04392882
Title: Effects of Legumes Consumption on Weight Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jong Ho Lee, Professor, Principal Investigator, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Legumes_Weight Reduction
Record Dates: First submitted 2020-05-06; First posted 2020-05-19 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Obese
Keywords: legumes; obesity; body weight; adiponectin; 8-epi-PGF2α; insulin resistance
MeSH Terms: conditions — Obesity; Body Weight; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Legume enriched diet group (Experimental): * Replacing 1/3 refined rice intake with legumes three times per day
  * Vegetable intake at least six units (30-70 g/unit) per day for sufficient dietary fiber intake
  * Regular 30-min walk after dinner each day
  Interventions: Behavioral: Legume enriched diet group
- Usual diet group (No Intervention): * Maintaining usual diet
  * Vegetable intake at least six units (30-70 g/unit) per day for sufficient dietary fiber intake
  * Regular 30-min walk after dinner each day

INTERVENTIONS:
Behavioral: Legume enriched diet group — * Replacing 1/3 refined rice intake with legumes three times per day
  * Vegetable intake at least six units (30-70 g/unit) per day for sufficient dietary fiber intake
  * Regular 30-min walk after dinner each day
  Arms: Legume enriched diet group

SUMMARY:
This is a 12-week, randomized nutritional intervention study to determine the effect of legumes consumption on body weight in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female volunteers between the ages of 20 to 70 years
2. Body mass index (BMI) of 25 kg/m2 or higher (based on Asia-Pacific guideline)
3. Volunteers who have agreed to participate in the study and provided a written content by him/herself

Exclusion Criteria:

1. Those with type 2 diabetes, cardiovascular disease, psychiatric problems, thyroid disorders, liver or kidney disease
2. Those under the use of any medications (antihypertensive, lipid-lowering, antiplatelet, antidiabetic, etc.).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2013-03-31 (Actual); Study Completion 2013-03-31 (Actual)

PRIMARY OUTCOMES:
Changes of BMI | 12 weeks
  Changes of weight in kilograms was assessed before and after the intervention.
  Changes of height in meters was assessed before and after the intervention.
  Weight and height were combined to report BMI in kg/m^2.
Changes of Insulin Resistance (IR) | 12 weeks
  Changes of fasting serum glucose in mmol/L was assessed before and after the intervention.
  Changes of fasting insulin in μIU/mL was assessed before and after the intervention.
  Fasting insulin and fasting glucose were combined to report IR using the following equation: homeostasis model assessment (HOMA)-IR=[fasting insulin (μIU/mL)×fasting glucose (mmol/L)] /22.5.
Changes of lipid profiles | 12 weeks
  Triglyceride in mg/dL was assessed before and after the intervention.
  Total-cholesterol in mg/dL was assessed before and after the intervention.
  HDL-cholesterol in mg/dL was assessed before and after the intervention.
  LDL-cholesterol was indirectly estimated using the friedewald formula: LDL-cholesterol= total-cholesterol-[HDL-cholesterol+(triglycerides/5)].
Changes of serum high C-reactive | 12 weeks
  Changes of serum high C-reactive in mg/L was assessed before and after the intervention.
Changes of urinary 8-epi-PGF2α | 12 weeks
  Changes of urinary 8-epi-PGF2α in pg/mg creatinine was assessed before and after the intervention.
Changes of adiponectin | 12 weeks
  Changes of adiponectin in ng/mL was assessed before and after the intervention.

IPD SHARING:
Plan to Share IPD: No